CLINICAL TRIAL: NCT04214821
Title: The Pharmacokinetics of Topical Levofloxacin 1.5% vs Topical Moxifloxacin 0.5%
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wan Haslina Wan Abdul Halim, Consultant Ophthalmologist-Cornea And Anterior Segment, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FF-2019-315
Record Dates: First submitted 2019-12-10; First posted 2020-01-02 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2019-12

CONDITIONS: Endophthalmitis
Keywords: Pharmacokinetic; Levofloxacin 1.5%; Moxifloxacin 0.5%
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Intervention Model Description: The qualified patients will be randomized on a 1:1 ratio into each treatment arm. Qualified eyes were further randomized into one of four subgroups, which specified the time between the last drop of study medication and the time of aqueous and vitreous humor sample collection (i.e., 1-, 2-, 4-, and 6-hour subgroups- about 32 patients per subgroup. Within each subgroups, there will be 16 of Levofloxacin group and 16 of Moxifloxacin group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Levofloxacin -1 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 1-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Levofloxacin Ophthalmic Solution
- Levofloxacin-2 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 2-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Levofloxacin Ophthalmic Solution
- Levofloxacin-4 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 4-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Levofloxacin Ophthalmic Solution
- Levofloxacin-6 hour group (Active Comparator): Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 6-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection
  Interventions: Drug: Levofloxacin Ophthalmic Solution
- Moxifloxacin-1 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 1-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution
- Moxifloxacin-2 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 2-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution
- Moxifloxacin-4 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 4-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution
- Moxifloxacin-6 hour group (Active Comparator): Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily (8am, 12pm, 4pm, 8pm) for 3 days prior to the surgery. On the day of surgery, there will be 6-hour gap between last drop of study medication and the time of aqueous and vitreous humor sample collection.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution

INTERVENTIONS:
Drug: Levofloxacin Ophthalmic Solution — Levofloxacin hydrate, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily for 3 days pre-operatively and one drop on the day of operation.
  Other Names: Cravit 1.5%
  Arms: Levofloxacin -1 hour group; Levofloxacin-2 hour group; Levofloxacin-4 hour group; Levofloxacin-6 hour group
Drug: Moxifloxacin Ophthalmic Solution — Moxifloxacin hydrochloride, an aqueous ophthalmic solution, to be given one drop at a time, 4 times daily for 3 days pre-operatively and one drop on the day of operation.
  Other Names: Vigamox 0.5%
  Arms: Moxifloxacin-1 hour group; Moxifloxacin-2 hour group; Moxifloxacin-4 hour group; Moxifloxacin-6 hour group

SUMMARY:
Endophthalmitis is defined as intraocular inflammatory disorder affecting the vitreous cavity that can result from exogenous or endogenous spread of infecting organisms into the eye. Patients presents with reduced or blurred vision, red eye, pain, and lid swelling. Endophthalmitis can progress into panophthalmitis, corneal infiltration and perforation, and finally phthisis bulbi. For exogenous endopthalmitis, the intraocular inflammation occurs due to a breach of the ocular compartment. The infectious agent indirectly introduced into the eye. This usually happens after intraocular surgery such as cataract surgery, vitrectomy, glaucoma filtration surgery, intravitreal injections, and other causes include penetrating ocular trauma or from adjacent periocular tissue. Several prophylactic measures have been taken to reduce the incidence of post-operative endopthalmitis post-cataract surgery, this includes the use of pre-operative topical levofloxacin, intracameral cefuroxime, and providone iodine as ocular surface preparation.The proposed study is to evaluate the pharmacokinetic parameters of Levofloxacin 1.5% vs Moxifloxacin 0.5% aqueous and vitreous fluid after topical administration on the anterior segment parameters.

DETAILED DESCRIPTION:
This is a prospective, double - blinded randomized clinical trial conducted in University Kebangsaan Malaysia Medical Centre (UKMMC) where there are two intervention arms. All patients from Ophthalmology Clinic in UKM Medical Centre from September 2019 till December 2021 will be involved in this study. Patients who fulfill the inclusion criteria will be included in this study. All eligible subjects will be asked to sign an informed consent.

The qualified patients will be randomized on a 1:1 ratio into each treatment arm. Qualified eyes were further randomized into one of four subgroups, which specified the time between the last drop of study medication and the time of aqueous and vitreous humor sample collection (i.e., 1-, 2-, 4-, and 6-hour subgroups- about 32 patients per subgroup-: 16 Levofloxacin, 16 Moxifloxacin.

For 3 days prior to the day of the elective vitrectomy surgery, subjects will instill exactly one drop of study medication into their operative eye four times daily. On the day of surgery (visit 2, day 4), patients will receive their final drop of study medication administered by trained study personnel at the study site.

Samples of aqueous (0.1 ml), and vitreous (0.2 ml) humour were taken simultaneously from the same patient at the commencement of surgery by paracentesis using a 30-gauge needle on a tuberculin syringe. All samples will be stored at -80°C as soon as possible until the concentrations of the drug will be measured.

Measurements for moxifloxacin and levofloxacin concentrations in aqueous fluid will be determined using HPLC with UV detection, which is currently undergoing method development and validation at the Faculty of Pharmacy, UKM. Measurements for moxifloxacin and levofloxacin concentrations in vitreous fluid will be outsourced to a laboratory at the Centre for Research and Instrument Management (CRIM) in UKM, due to the high sensitivity required to determine the drugs' concentrations in vitreous fluid.

A compartmental analysis will be carried out using AUC0-6, Cmax, and time to Cmax (Tmax) will be determined by direct observation. The median AUC0-6 calculation will be performed using the linear trapezoid method. A Kruskal-Wallis nonparametric one-way analysis of variance (ANOVA) will be used to detect differences between the concentrations in each treatment arm at various time points. A p value of <0.05 is considered statistically significant. Data management and statistical analysis will be performed using the PKNCA package in R and SPSS ver 23.0, whichever deemed suitable.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for vitrectomy for macula hole , ERM, RD surgery
* Age 18 and above
* Not on any topical medication

Exclusion Criteria:

* Patients with underlying ocular surface disease
* Fluoroquinolone allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of volume of distribution (Maximum Plasma Concentration) of Levofloxacin 1.5% vs Moxifloxacin 0.5% in the aqueous and vitreous fluid. | Throughout study completion, an average of 2 years
  A compartmental analysis will be carried out. Data for the pooled aqueous and vitreous humor concentrations in each of the treatment groups, n, mean, SD, median, and coefficient of variation, and range values for each time point will be calculated. Since each patient contributed to this pooled non-compartmental analysis at a specified time point, Maximum Plasma Concentration (Cmax), and time to Cmax (Tmax) will be determined by direct observation.
Comparison of volume of distribution (Area under the plasma concentration versus time curve) of Levofloxacin 1.5% vs Moxifloxacin 0.5% in the aqueous and vitreous fluid. | Throughout study completion, an average of 2 years
  A compartmental analysis will be carried out. Data for the pooled aqueous and vitreous humor concentrations in each of the treatment groups, n, mean, SD, median, and coefficient of variation, and range values for each time point will be calculated. Since each patient contributed to this pooled non-compartmental analysis at a specified time point, a representative Area under the plasma concentration versus time curve (AUC0-6) will be determined by direct observation. The median AUC0-6 calculation will be performed using the linear trapezoid method.
Comparison of concentration of Levofloxacin 1.5% and Moxifloxacin 0.5% in the aqueous and vitreous fluid. | Throughout study completion, an average of 2 years
  The mean concentration vs time of last drop (i.e. AUC) will be plotted for both levofloxacin 1.5% and moxofloxacin 0.5% in aqueous and vitreous fluids. A Kruskal-Wallis non-parametric one-way analysis of variance (ANOVA) will be used to detect differences between the concentrations in each treatment arm at various time points.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Haslina Wan Abdul Halim, M.D, Study Chair — Department of Ophthalmology, UKM Medical Centre
Locations (2):
- Malaysia (2):
  - UKM Medical Centre, Cheras, Kuala Lumpur
  - Faculty of Pharmacy, National University of Malaysia, Kuala Lumpur, Kuala Lumpur

REFERENCES:
- [Background] Jackson TL, Paraskevopoulos T, Georgalas I. Systematic review of 342 cases of endogenous bacterial endophthalmitis. Surv Ophthalmol. 2014 Nov-Dec;59(6):627-35. doi: 10.1016/j.survophthal.2014.06.002. Epub 2014 Jun 18. PMID 25113611
- [Background] Nishida T, Ishida K, Niwa Y, Kawakami H, Mochizuki K, Ohkusu K. An eleven-year retrospective study of endogenous bacterial endophthalmitis. J Ophthalmol. 2015;2015:261310. doi: 10.1155/2015/261310. Epub 2015 Jan 31. PMID 25802752
- [Background] Kernt M, Kampik A. Endophthalmitis: Pathogenesis, clinical presentation, management, and perspectives. Clin Ophthalmol. 2010 Mar 24;4:121-35. doi: 10.2147/opth.s6461. PMID 20390032
- [Background] Puustjarvi T, Terasvirta M, Nurmenniemi P, Lokkila J, Uusitalo H. Penetration of topically applied levofloxacin 0.5% and ofloxacin 0.3% into the vitreous of the non-inflamed human eye. Graefes Arch Clin Exp Ophthalmol. 2006 Dec;244(12):1633-7. doi: 10.1007/s00417-006-0360-0. PMID 16715252
- [Result] Results of the Endophthalmitis Vitrectomy Study. A randomized trial of immediate vitrectomy and of intravenous antibiotics for the treatment of postoperative bacterial endophthalmitis. Endophthalmitis Vitrectomy Study Group. Arch Ophthalmol. 1995 Dec;113(12):1479-96. PMID 7487614
- [Result] Hariprasad SM, Blinder KJ, Shah GK, Apte RS, Rosenblatt B, Holekamp NM, Thomas MA, Mieler WF, Chi J, Prince RA. Penetration pharmacokinetics of topically administered 0.5% moxifloxacin ophthalmic solution in human aqueous and vitreous. Arch Ophthalmol. 2005 Jan;123(1):39-44. doi: 10.1001/archopht.123.1.39. PMID 15642810
- [Result] Robertson SM, Curtis MA, Schlech BA, Rusinko A, Owen GR, Dembinska O, Liao J, Dahlin DC. Ocular pharmacokinetics of moxifloxacin after topical treatment of animals and humans. Surv Ophthalmol. 2005 Nov;50 Suppl 1:S32-45. doi: 10.1016/j.survophthal.2005.07.001. PMID 16257309
- [Result] Bucci FA Jr, Nguimfack IT, Fluet AT. Pharmacokinetics and aqueous humor penetration of levofloxacin 1.5% and moxifloxacin 0.5% in patients undergoing cataract surgery. Clin Ophthalmol. 2016 May 2;10:783-9. doi: 10.2147/OPTH.S91286. eCollection 2016. PMID 27194905
- [Result] Jackson MA, Schutze GE; COMMITTEE ON INFECTIOUS DISEASES. The Use of Systemic and Topical Fluoroquinolones. Pediatrics. 2016 Nov;138(5):e20162706. doi: 10.1542/peds.2016-2706. PMID 27940800
- [Result] Watanabe R, Nakazawa T, Yokokura S, Kubota A, Kubota H, Nishida K. Fluoroquinolone antibacterial eye drops: effects on normal human corneal epithelium, stroma, and endothelium. Clin Ophthalmol. 2010 Oct 21;4:1181-7. doi: 10.2147/OPTH.S13672. PMID 21060669
- [Result] Hanscom TA. Postoperative endophthalmitis. Clin Infect Dis. 2004 Feb 15;38(4):542-6. doi: 10.1086/381262. Epub 2004 Jan 26. PMID 14765348